CLINICAL TRIAL: NCT06246487
Title: Assessing Heterogeneity of Treatment Response in Children With Autism Spectrum Disorder
Brief Title: Sensory Intervention for Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB202200163; W81XWH-21-1-0594 (Other Grant/Funding Number: US Dept of Defense)
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Occupational Therapy Intervention
  Interventions: Behavioral: Occupational Therapy Intervention
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Occupational Therapy Intervention — Children randomized to the intervention condition will receive a sensory enriched intervention 2x's per week, 60-minutes per session, for 16 weeks. The intervention will follow a codified protocol developed by Dr. Bodison that is theoretically grounded in neurodevelopmental research. The interveners will be occupational therapists who will be trained by Dr. Bodison to deliver the codified, intervention protocol to provide a personally customized set of therapeutically guided environmental interactions. Because, at its core, the intervention emphasizes playful interaction with a sensory enriched environment, the intervention room will be equipped with swings, scooter boards, climbing equipment, bolsters, and large carpeted barrels. Within this setting, using the codified manual of intervention developed by Dr. Bodison, the intervener will structure activities to provide tactile and proprioceptive input to address the child's individualized areas of need.
  Arms: Intervention

SUMMARY:
Greater than 80% of children with autism spectrum disorder (ASD) experience sensory differences that make it difficult for them to fully participate in meaningful everyday activities. In this research study, we will use MRI and behavioral methods to assess how sensory interventions might change sensory brain structures, allowing us to better predict which sensory interventions might work best for whom.

ELIGIBILITY:
Inclusion Criteria: Male children 6 years, 0 months to 8 years, 6 months of age with a diagnosis of autism spectrum disorder (ASD) will qualify for inclusion. Our inclusion age ensures all study participants will complete intervention/control conditions and be retested before they turn 9 years of age. Additional inclusion criteria include:

1. The families of children will have access to transportation to attend intervention sessions 2 times per week for 16-weeks.
2. Children who qualify will be verbal, and will speak and understand English. The native language of caregivers can include Spanish.
3. Children who qualify will have sensorimotor delays as assessed by the study team using the standardized, norm-referenced assessments described in this research proposal (z-scores on 3 of 5 tests -1.0 or lower).

Exclusion Criteria: Children younger than 6 years of age or older than 8 years, 6 months of age will be excluded. Additional exclusion criteria include:

1. Female children
2. Auditory hyperresponsivity as assessed during screening procedures.
3. Medical co-morbidities such as extreme prematurity (less than 28 weeks), blindness, deafness, cerebral palsy, Down Syndrome, tuberous sclerosis, or head-injury with loss of consciousness.
4. History of individual occupational therapy services in a clinical setting that includes sensory equipment.
5. Non-removable metal in the head or body (e.g. dental fillings & braces, metal pins, screws or plates).
6. Children unable to complete neurocognitive or sensorimotor testing.
7. Children unsuccessful in 3 mock scanning sessions during baseline testing.

Ages: 6 Years to 9 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Neuroimaging | 16 weeks
  Pre vs, post magnetic resonance imaging scans

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-03-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT06246487/ICF_000.pdf